CLINICAL TRIAL: NCT02007187
Title: A Randomized, Double-blind, Multicenter, Parallel Controlled Clinical Trial of Danhong Injection in the Treatment of Unstable Angina Pectoris
Brief Title: Danhong Injection in the Treatment of Unstable Angina Pectoris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: China Food and Drug Administration (Other Government)
Responsible Party: Principal Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011ZX09304-07V1.2
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Unstable Angina Pectoris
Keywords: Unstable Angina Pectoris; Randomized Controlled Trial; Traditional Chinese Medicine
MeSH Terms: conditions — Angina, Unstable | interventions — danhong

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Danhong injection (Experimental): Based on the standard medical care, 40ml of Danhong injection, added into 250ml of 0.9% saline, given by continuous IV infusion at 2.5ml/min within 2-3 hours every day for 7 days.
  Interventions: Drug: Danhong injection; Other: Standard medical care
- Placebo (Placebo Comparator): Based on the standard medical care, placebo was 40ml of 0.9% saline, added into 250ml of 0.9% saline, given by continuous IV infusion at 2.5ml/min within 2-3 hours every day for 7 days.
  Interventions: Other: Standard medical care; Drug: Placebo

INTERVENTIONS:
Drug: Danhong injection — A kind of injection made from two kind of Chinese herbs: salvia miltiorrhiza and safflower
  Arms: Danhong injection
Other: Standard medical care — Standard medical care is in accordance with China Guideline for the diagnosis and treatment of unstable angina (UA) and non-ST-elevation myocardial infarction (NSTEMI) (2007) issued by Chinese Society of Cardiology of Chinese Medical Association
Drug: Placebo — 0.9% saline added into 250ml 0.9% saline by an independent research nurse, sealed with brown bag in order to make the investigators and patients blinded, using brown infusion tube for infusion.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of Danhong injection in the treatment of unstable angina pectoris.

ELIGIBILITY:
Inclusion Criteria:

* Female or male inpatients.
* Age: 35 - 75 years.
* Patients with clinical diagnosis of unstable stable angina according to China Guideline for the diagnosis and treatment of unstable angina (UA) and non-ST-elevation myocardial infarction (NSTEMI) (2007) issued by Chinese Society of Cardiology of Chinese Medical Association, including one of the following conditions.
* Clinical diagnosis of "Xueyu Zheng" (Blood Stasis Syndrome) as the scores of Chinese medicine symptoms scales of "Xueyu Zheng" in UA ≥ 15. The Chinese medicine symptoms scales of "Xueyu Zheng" is a 6-item questionnaire including the symtoms as following: (1)chest pain-10, (2)chest distress-10, (3) palpitation-5, (4)purple or dark lip-5, (5) purple or dark tongue-5, (6) unsmooth pulse-5.
* Patient is willing to participate voluntarily and to sign a written patient informed consent.

Exclusion Criteria:

* Patients with severe heart failure (EF<35%);
* Patients with history of infection, fever, trauma, surgery(exclude PCI) and inflammation in the past month;
* Patients with active tuberculosis or rheumatological disorders;
* Patients with renal dysfunction (Male: CCr>2.5mg/dl; Female: CCr>2.0mg/dl);
* Patients with liver dysfunction (any value of serum aminotransferase more than triple normal value);
* Patients with history of hematopoietic system diseases;
* Patients with mental disorder;
* Patients with history of drug-induced bleeding or history of bleeding caused by warfarin;
* Patients with malignant tumor;
* Patients with history of organ transplant;
* Woman with pregnancy, lactation or positive result of pregnancy test;
* Patients who is participating in other trials or has been participated in other trials in recent 3 months;
* Patients who were unable to participate in the study as judged by investigator.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the Quantification score of angina pectoris at Day 7 | Day 7
  Quantification score of angina pectoris is a 4-item questionnaire that quantifies the frequency of angina, the duration of angina at every attack, the severity of angina and the use of nitroglycerin in a week. Scores range from 0 to 24; higher scores indicate worse health status.

SECONDARY OUTCOMES:
Total score of symptoms questionnaire of TCM | Day 0, Day 7
  The symptoms questionnaire of TCM consists of 6 symptoms that described in traditional Chinese medicine, including chest pain, chest distress, palpitation, dark-purple lip, dark-purple tongue and unsmooth pulse. Each symptom was assessed by the Visual Analogue Scale（VAS），where a higher score meant higher severity.
Use of Short-acting Nitrates | Day 0, Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 28
Change in the electrocardiogram (ECG) | Day 0, Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 28
  ECG will be done five times every day, when 5-10 min before use of nitrates or Danhong injection, 5-10 min after use of nitrates or Danhong injection, at the time 22:00. If there is an angina attack, an additional ECG should be done when the angina attacks.
The proportion of patients who are undergoing PCI | Day 7, Day 28
Change in Seattle Angina Questionnaire | Day 0, Day 28
  Seattle Angina Questionnaire, a 19-item questionnaire that quantifies physical limitations due to angina, any recent change in the severity of angina, the frequency of angina, satisfaction with treatment, and quality of life. Scores range from 0 to 100; higher scores indicate better health status.With a score of 20 or more on the angina-frequency scale indicating that the patient was clinically significant change.
Incidence of adverse events (including serious adverse events) in 28 days | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Wang, M.D., Ph.D., Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences; Xian Wang, M.D., Principal Investigator — Dongzhimen Hospital, Beijing; Xiao-xi Du, Professor, Study Director — China Food and Drug Administration
Locations (9):
- China (9):
  - Xuanwu Hospital, Beijing, Beijing Municipality
  - Dongzhimen Hospital affiliated to Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - The First Affiliated Hospital of Heilongjiang University of Traditional Chinese Medicine, Harbin, Heilongjiang
  - Zhengzhou No.7 People's Hospital, Zhengzhou, Henan
  - The First Hospital of Changsha, Changsha, Hunan
  - The Affiliated Hospital to Changchun University of Chinese Medicine, Changchun, Jilin
  - Hospital 463 of P.L.A., Shenyang, Liaoning
  - First Teaching Hospital of Tianjin University of T.C.M., Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Chen L, Fu G, Hua Q, Zhu HY, Deng Y, Wu W, Zhao YJ, Yang XY, Yang BS, Zhou YB, Liu J, Yu YN, Chen BW, Wang X, Wang Z. Efficacy of add-on Danhong injection in patients with unstable angina pectoris: A double-blind, randomized, placebo-controlled, multicenter clinical trial. J Ethnopharmacol. 2022 Feb 10;284:114794. doi: 10.1016/j.jep.2021.114794. Epub 2021 Oct 31. PMID 34732357